CLINICAL TRIAL: NCT02096185
Title: Is Any Additional Information Gained Regarding Lesion to Margin Measurement Using 3D Tomosynthesis Imaging Versus 2D Conventional Digital Imaging When Imaging Specimens of Breast Tissue Removed at Therapeutic Surgery
Brief Title: Is Any Additional Information Gained Regarding Margins Using 3D Tomosynthesis Vs 2D Conventional Digital Imaging When Imaging Operative Breast Specimens?
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Sandwell & West Birmingham Hospitals NHS Trust (Other)
Responsible Party: Principal Investigator, Jennifer Waldron, Consultant Radiographer, Sandwell & West Birmingham Hospitals NHS Trust
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Diagnostic
Other Study IDs: Breast Specimen Imaging Ver3
Record Dates: First submitted 2014-03-21; First posted 2014-03-26 (Estimated); Last update posted 2016-10-21 (Estimated); Status verified 2015-11

CONDITIONS: Breast Cancer
Keywords: Breast cancer; Surgery; Specimen imaging
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 3 dimensional tomosynthesis imaging (Experimental): Breast specimen to be x-rayed using both conditions 3 dimensional tomosynthesis imaging 2 dimensional conventional digital imaging
  Interventions: Radiation: 3 dimensional tomosynthesis imaging
- 2 dimensional digital imaging (Experimental): Breast specimens to be x-rayed under both conditions 3 dimensional tomosynthesis imaging 2 dimensional digital imaging
  Interventions: Radiation: 2 dimensional digital imaging

INTERVENTIONS:
Radiation: 3 dimensional tomosynthesis imaging — Each operative specimen will be imaged twice using each condition
  Arms: 3 dimensional tomosynthesis imaging
Radiation: 2 dimensional digital imaging
  Arms: 2 dimensional digital imaging

SUMMARY:
Patients who are diagnosed with breast cancer will have surgery to remove the tumour. Where this is a local excision not mastectomy, the tissue removed is sent for x-ray imaging to assess that the abnormality has been removed and give an estimation of the distance from lesion to specimen edge. This allows the surgeon to decide whether to remove more tissue or not at the time. This study is designed to compare whether more accurate information about lesion to margin measurement can be obtained using 3 dimensional tomosynthesis imaging compared to 2 dimensional conventional digital imaging which is the type of imaging currently used. This has the potential to prevent some patients requiring a second operation to remove more tissue if the margins of the specimen are still involved with tumour.

The study involves x-raying the specimen under both conditions when it arrives from theatre. Only the 2D image will be reviewed at the time as is current practice. The 3D image will be reviewed later and the measurements for lesion to specimen margin compared. The lesion to margin measurement as recorded by the pathologist will be taken as the 'gold standard' and the imaging measurements will also be compared to that.

In theory, the use of 3D tomosynthesis should allow more accurate lesion to margin measurement because 3D can provide better visualisation of the lesion edges by removing the effect of superimposed tissue.

The hypothesis states that the use of 3 dimensional tomosynthesis imaging should provide better lesion visualisation compared to 2 dimensional conventional digital imaging thus allowing more accurate lesion to margin measurement.

ELIGIBILITY:
Inclusion Criteria:

* Patient requires surgery to remove breast cancer and operative specimen needs to be x-rayed

Exclusion Criteria:

* Patients with breast cancer who need mastectomy

Min Age: 30 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2014-05; Primary Completion 2017-04 (Estimated); Study Completion 2017-05 (Estimated)

PRIMARY OUTCOMES:
Shortest distance in mm from visible lesion to specimen margin | 1 year
  2D conventional digital imaging - measured at time of surgery and info relayed to surgeon in theatre 3D tomosynthesis imaging - measured later with operator blinded to the 2D measurement Pathological measurement - final measurement used as the 'gold standard'

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Waldron, Principal Investigator — Sandwell & West Birmingham Hospitals NHS Trust
Locations (1):
- Sandwell and West Birmingham Hospitals NHS Trust, Birmingham, West Midlands, United Kingdom